CLINICAL TRIAL: NCT06795685
Title: The Role of Pre-natal Ultrasound in Predicting Outcomes of Fetal Ovarian Cysts
Acronym: OVARY22
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: OVARY 22
Record Dates: First submitted 2024-12-03; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-10

CONDITIONS: Fetal Ovarian Cyst
Keywords: ultrasound
MeSH Terms: conditions — Neonatal ovarian cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate whether there are any prenatal ultrasound features that may predict the need for postnatal surgery versus spontaneous regression of such formations, so that better counseling can be provided to parents even in the prenatal period.

DETAILED DESCRIPTION:
The rationale of the study is to define the role of prenatal ultrasonography in diagnostic framing and prognostic guidance in cases of suspected fetal ovarian cyst detection. Prenatal ultrasonography in such cases detects the presence of a pelvic formation in female fetuses, although the differential diagnosis is not always straightforward and can only be placed with certainty in the postnatal period. The investigators will therefore retrospectively assess postnatal outcomes in newborns prenatally diagnosed with ovarian cysts and investigate the presence of any prenatal ultrasound findings most associated with an unfavorable postnatal prognosis in terms of need for surgery and fetal complications. This will allow the investigators to more precisely delineate the timing of serious prenatal ultrasound checks once the diagnosis of fetal ovarian cyst is established.

Ultrasound follow-up has been performed in all infants with prenatal ultrasound suspicion of ovarian cyst and continues until the cyst disappears, which occurs on average within the first six to 12 months of life. Follow-up therefore is generally 12 months, but may be discontinued early in case of earlier resolution of the cyst.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* Age greater than or equal to 18 years
* Detection of suspected fetal ovarian cyst on ultrasonography
* Performance of delivery at the division of Obstetrics and Prenatal Age Medicine

Exclusion Criteria:

None

Ages: 18 Years to 44 Years | Sex: Female
Age Groups: Adult
Study Population: Patients who were evaluated with serial ultrasound checks at the outpatient clinics of the division of Obstetrics and Prenatal Age Medicine of IRCCS Azienda Ospedaliero Universitaria di Bologna, Policlinico di Sant'Orsola for the presence of suspected fetal ovarian cyst diagnosis between 2008 and 2021 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Association between ovarian cyst characteristics and the performance of cyst excision surgery on the newborn. | Up to 100 weeks
  The outcome of the primary aim will be the percentage of infants who underwent surgery vs those in whom the formation went into spontaneous regression

SECONDARY OUTCOMES:
Postnatal Outcomes | Up to 100 weeks
  Description of the cohort of fetuses prenatally diagnosed with suspected ovarian cyst
Changes in the ultrasonographic features of the cyst in the prenatal period | up to 100 weeks
  Description of the cohort of fetuses prenatally diagnosed with suspected ovarian cyst
Type of cyst on histologic examination in case of surgery | Up to 100 weeks
  - mode and type of surgery
  Description of the cohort of fetuses prenatally diagnosed with suspected ovarian cyst
Mode and type of surgery | Up to 100 weeks
  Description of the cohort of fetuses prenatally diagnosed with suspected ovarian cyst

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Montaguti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy